CLINICAL TRIAL: NCT04814797
Title: The Study of Capnography for the Follow-up of Cystic Fibrosis Children With or Without Gas Trapping
Brief Title: Use of Capnography for the Follow-up of Cystic Fibrosis Children
Acronym: MUCOCAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr. Iulia IOAN, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI150
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
Keywords: Pulmonary function testing
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CF children "with gas trapping": CF children "with gas trapping" will be defined by a ratio between the difference of functional residual capacity (FRC) obtained by plethysmography (FRCpleth) and FRC obtained by helium dilution method (FRCHe) divided by the FRCpleth of >10%
  Interventions: Other: Capnography data included in Lung Clearance Index measurement
- CF children "without gas trapping": CF children "without gas trapping" will be defined by a ratio between the difference of the functional residual capacity (FRC) obtained by plethysmography (FRCpleth) and FRC obtained by helium dilution method (FRCHe) divided by the FRCpleth of ≤10%
  Interventions: Other: Capnography data included in Lung Clearance Index measurement

INTERVENTIONS:
Other: Capnography data included in Lung Clearance Index measurement — Capnography data included in Lung Clearance Index measurement (a pulmonary function test included in routinely yearly follow-up of cystic fibrosis children) will be collected and analyzed

SUMMARY:
The respiratory system involvement in cystic fibrosis(CF) influences the prognosis and course of disease. Respiratory assessment is based on spirometry, but its main parameter, the maximal expiratory volume in the first second (FEV1), does not reflect the initial peripheral impairment of airways. Another pulmonary function test (PFT) validated for CF children follow-up is measurement of "gas trapping", reflecting ventilation inhomogeneity and incipient airways impairment. "Gas trapping" can be obtained by lung volume measurement (functional residual capacity, FRC) by plethysmography and helium dilution technique, but these tests are inconvenient for children due to their long length (~30min). A complete PFT is routinely performed once a year. It also includes a measurement of Lung Clearance Index (LCI) reflecting ventilation inhomogeneity. Capnography is a non-invasive PFT technique, does not require subject's active cooperation, is of short duration and could replace the traditional PFT for CF children follow-up. The capnograph is integrated into the device measuring LCI and data can be retrieved and analyzed afterwards. Capnographic indices reflect ventilation inhomogeneity.

The hypothesis is that capnographic indices change in the presence/absence of "gas trapping" in CF children.

The main objective is to show that the capnographic index of efficacy (EFFi) is significantly different between CF children "with gas trapping" and CF children "without gas trapping". The secondary objectives are:

* to compare the other capnographic indices between CF children "with gas trapping" and CF children "without gas trapping": the slope of the ascending phase, α; the slope of the alveolar plateau, β; the angle Q between α and β; the positive peak of the first-order derivative, F'CO2, which reflects the ascending phase; the first negative peak of the 2nd order derivative, F "CO2, which reflects the curvature between the ascending phase and the alveolar plateau.
* to compare the results of the capnographic indices with the results of the FEV1 in identifying the presence / absence of "gas trapping";
* to compare the results of the capnographic indices with the results of the LCI in identifying the presence / absence of "gas trapping"

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common inherited genetic disorder in Caucasian children. It affects several organs, the most important being the involvement of the respiratory system. The respiratory condition influences the prognosis and the course of the disease, the respiratory complications being the main cause of mortality and morbidity. The respiratory assessment is based on spirometry, but the maximal expiratory volume in the first second (FEV1) does not reflect the initial peripheral impairment of airways and can remain within normal limits for a long time. Another pulmonary function test (PFT) validated for the follow-up of CF children is the measurement of "gas trapping", very frequent in these children, reflecting the ventilation inhomogeneity and incipient airways impairment. "Gas trapping" can be obtained by the measurement of lung volume (functional residual capacity, FRC) by plethysmography and helium dilution technique, but these tests are very inconvenient for children due to their long length (~ 30 minutes). This complete PFT is routinely performed every year. It also includes a measurement of Lung Clearance Index (LCI) which reflects the presence of ventilation inhomogeneity. Capnography is a non-invasive PFT technique that does not require subject's active cooperation, is of short duration and could replace the traditional PFT techniques for the follow-up of CF children. Capnographic indices also reflect the presence of ventilation inhomogeneity. The capnograph is integrated into the device that measures the LCI and data can be retrieved and analyzed following the LCI measurement.

In this study, 2 groups of children will be identified by the gold-standard: 1 / children with "gas trapping" (defined by the ratio between the difference in the plethysmographic FRC (FRCpleth) and FRC obtained by the helium dilution technique (FRCHe) divided by FRCpleth of >10%) and 2 / children without "gas trapping" (defined by (FRCpleth-FRCHe) / FRCpleth of ≤ <10%). Capnography data (included in LCI measurement) will be collected in these children and capnographic indices will be compared between these two groups.

The study hypothesis is that capnographic indices change in the presence or absence of "gas trapping" in CF children.

The importance of capnography is that is a test less inconvenient for follow-up and better accepted by children because of its short length, easy-to-use tool for monitoring disease progression and monitoring the effectiveness of treatments.

The main objective is to show that the capnographic index of efficacy (EFFi), in CF children is significantly different between subjects "with gas trapping" (defined by the gold standard ((FRCpleth - FRCHe) / FRCpleth) > 10%) and subjects "without gas trapping" (defined by the gold standard ((FRCpleth-FRCHe) / FRCpleth) ≤10%).

The secondary objectives are:

* to compare the other capnographic indices between CF children "with gas trapping" and CF children "without gas trapping": the slope of the ascending phase, α; the slope of the alveolar plateau, β; the angle Q between α and β; the positive peak of the first-order derivative, F'CO2, which reflects the ascending phase; the first negative peak of the 2nd order derivative, F"CO2, which reflects the curvature between the ascending phase and the alveolar plateau.
* to compare the results of the capnographic indices with the results of the FEV1 in identifying the presence / absence of "gas trapping";
* to compare the results of the capnographic indices with the results of the LCI in identifying the presence / absence of "gas trapping",

ELIGIBILITY:
Inclusion Criteria: common to the 2 groups studied are as follows:

* child aged 6 to 17 inclusive;
* child diagnosed with cystic fibrosis (CF) and follow-up at the pediatric reference center of University Children's Hospitals of Nancy and Trousseau Hospital in Paris
* child for whom data from a complete routinely pulmonary function testing are available
* child who did not object to his/her participation
* child whose parental authority have received full information on the current research and have not objected to the participation of their child

The criterion for inclusion in the group "with gas trapping" is gold standard (FRCpleth-FRCHe) / FRCpleth> 10% The criterion for inclusion in the group "without gas trapping" is gold standard (FRCpleth-FRCHe) / FRCpleth ≤10%

The number of subjects potentially recruited "with gas trapping" and "without gas trapping" is unbalanced (imbalance estimated at ½ and taken into account in the calculation of the number of subjects required). In order not to go beyond this imbalance, recruitment in one of the two groups (instruction applied by center) will be stopped as soon as this group has reached the planned number of subjects and will continue only with the inclusion of subjects in the other group.

Exclusion Criteria:

* other chronic respiratory pathology (bronchopulmonary dysplasia, virosis sequelae, inhalation pathology, thoraco-pulmonary malformation, tracheomalacia);
* anatomical or functional abnormalities of the pharyngolaryngeal pathway (tonsils hypertrophy grade 3 or 4, laryngomalacia, subglottic stenosis, vocal cord paralysis, any other laryngeal obstacle);
* congenital or acquired heart disease.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children are recruited from subjects diagnosed with cystic fibrosis followed-up at the pediatric reference center of University Children's Hospital of Nancy and Trousseau of Paris (46 children from Nancy and 30 children from Paris). These children are referred by the pneumopediatricians to the Pediatric Pulmonary Function Testing Lab for a complete, annually, routinely follow-up assessment of respiratory function.
  An analysis of the capnography data included in the Lung Clearance Index measurement, which is part of the routine assessment of the CF child, will be performed.
  The complete routine yearly PFT in order to ensure the follow-up in CF children is composed of 4 techniques: measurement of lung volumes by plethysmography (1), measurement of lung volumes by helium dilution technique (2); LCI measurement (3); spirometry (4). The outcomes needed for this research are obtained by these techniques.
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficiency index (EFFi) Gold standard (CRFpleth - CRFHe) / CRFpleth to differentiate between subjects "with" gas trapping (defined by> 10%) and subjects "without" gas trapping (defined by ≤10%). | through study completion, an average of 6 months
  Value of the capnographic efficiency index (EFFi), for each of the children of the two groups studied . easurement included in the device that measures LCI, collected after LCI measurement

SECONDARY OUTCOMES:
Other capnographic indices | through study completion, an average of 6 months
  Value of capnographic indices for each of the children of the two groups studied ; Data collected after PFT
Forced expiratory volume in the first second (FEV1) | through study completion, an average of 6 months
  The value of FEV1 obtained by spirometry for each of the children of the two groups studied
Lung Clearance Index (LCI) | through study completion, an average of 6 months
  Value of Lung Clearance Index for each of the children of the two groups studied

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de NANCY, Nancy
  - Hôpital ARMAND TROUSSEAU, Paris

REFERENCES:
- [Background] Robinson PD, Latzin P, Ramsey KA, Stanojevic S, Aurora P, Davis SD, Gappa M, Hall GL, Horsley A, Jensen R, Lum S, Milla C, Nielsen KG, Pittman JE, Rosenfeld M, Singer F, Subbarao P, Gustafsson PM, Ratjen F; ATS Assembly on Pediatrics. Preschool Multiple-Breath Washout Testing. An Official American Thoracic Society Technical Statement. Am J Respir Crit Care Med. 2018 Mar 1;197(5):e1-e19. doi: 10.1164/rccm.201801-0074ST. PMID 29493315
- [Background] BEDELL GN, MARSHALL R, DUBOIS AB, COMROE JH. Plethysmographic determination of the volume of gas trapped in the lungs. J Clin Invest. 1956 Jun;35(6):664-70. doi: 10.1172/JCI103323. No abstract available. PMID 13319505
- [Background] Kraemer R, Schoni MH. Ventilatory inequalities, pulmonary function and blood oxygenation in advanced states of cystic fibrosis. Respiration. 1990;57(5):318-24. doi: 10.1159/000195864. PMID 2284509
- [Background] O'Donnell CR, Bankier AA, Stiebellehner L, Reilly JJ, Brown R, Loring SH. Comparison of plethysmographic and helium dilution lung volumes: which is best for COPD? Chest. 2010 May;137(5):1108-15. doi: 10.1378/chest.09-1504. Epub 2009 Dec 18. PMID 20022972
- [Background] Jarenback L, Tufvesson E, Ankerst J, Bjermer L, Jonson B. The Efficiency Index (EFFi), based on volumetric capnography, may allow for simple diagnosis and grading of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Jun 27;13:2033-2039. doi: 10.2147/COPD.S161345. eCollection 2018. PMID 29988757
- [Background] Ioan I, Demoulin B, Duvivier C, Leblanc AL, Bonabel C, Marchal F, Schweitzer C, Varechova S. Frequency dependence of capnography in anesthetized rabbits. Respir Physiol Neurobiol. 2014 Jan 1;190:14-9. doi: 10.1016/j.resp.2013.09.002. Epub 2013 Sep 12. PMID 24035836
- [Background] Gustafsson PM, Aurora P, Lindblad A. Evaluation of ventilation maldistribution as an early indicator of lung disease in children with cystic fibrosis. Eur Respir J. 2003 Dec;22(6):972-9. doi: 10.1183/09031936.03.00049502. PMID 14680088
- [Background] You B, Peslin R, Duvivier C, Vu VD, Grilliat JP. Expiratory capnography in asthma: evaluation of various shape indices. Eur Respir J. 1994 Feb;7(2):318-23. doi: 10.1183/09031936.94.07020318. PMID 8162985